CLINICAL TRIAL: NCT04109157
Title: Test-retest Reliability of 20-minute Pad Test Infused With Strong-desire Amount of Water In Bladder in Women With Urodynamic Stress Incontinence
Brief Title: Test-retest Reliability of 20-minute Pad Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200612063R
Record Dates: First submitted 2019-09-23; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-08

CONDITIONS: Urodynamic Stress Incontinence
Keywords: Pad test; Test-retest reliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study population (Other): Women who had fulfilled the standardization of terminology of lower urinary function from ICS were diagnosed as urodynamic stress incontinence (USI) after urodynamic study (UDS) and enrolled for analysis in this study.
  Interventions: Diagnostic Test: 20-minute pad test

INTERVENTIONS:
Diagnostic Test: 20-minute pad test — Our 20-minute modified pad test was described previously proposed first by Hahn and Fall and modified by Sand and Ostergard. Each patient's bladder was emptied with a transurethral catheter and filled to the SD amount of sterile water for test. The catheter was removed, and then the patient returned to a standing position with a pre-weighed perineal pad placed on the underwear. The patient was asked to cough 10 times, bear down 10 times, do 10 deep knee bends, jump up and down on the spot 10 times, wash her hands under cold water for 1 minute, walk up and down five stairs 10 times, walk in the hall for 10 minute, and then return for removal of the pad. The pad was then weighed and the net weight was calculated by subtracting from the original dry weight to achieve a measure of the total urine loss during the 20 minute exercise. The pad weight was measured in grams and the accuracy of the scale was 1 gram. The positive pad weight result was defined as more than 1 gram of leakage.

SUMMARY:
In our department, we performed a 20-minute pad test since 2005. The 20-minute pad test uses 250 mL of sterile water instilled directly into an empty bladder with a catheter rather than relying on walking for 30 minutes at the beginning of a one-hour pad test. We previously reported that 20-minute pad test has better sensitivity than the one-hour pad test in women with stress urinary incontinence (SUI). Due to the different bladder capacity in each patient, we tried to infuse strong-desire (SD) amounts of water that can more precisely reflect the full bladder capacity in each patient. We found an even better sensitivity when the 20-minute pad test was infused with SD amount of water in women with SUI compared with infusion with 250 mL of water in the bladder.

As to short-term pad test, previous studies had some concerned about the reliability and reproducibility. Thus, undertaking our previous two studies, we want to evaluate the test-retest reliability of the 20-minute pad test infused with SD amount of water in bladder in women with SUI.

DETAILED DESCRIPTION:
Between August 2007 and December 2010, a total of 89 women with SUI were recruited. Of them, 67 (75%) women who had fulfilled the standardization of terminology of lower urinary function from ICS were diagnosed as urodynamic stress incontinence (USI) after urodynamic study (UDS) and enrolled for analysis in this study. Our 20-minute modified pad test was described previously proposed first by Hahn and Fall and modified by Sand and Ostergard. Each patient's bladder was emptied with a transurethral catheter and filled to the SD amount of sterile water for test. The catheter was removed, and then the patient returned to a standing position with a pre-weighed perineal pad placed on the underwear. The patient was asked to cough 10 times, bear down 10 times, do 10 deep knee bends, jump up and down on the spot 10 times, wash her hands under cold water for 1 minute, walk up and down five stairs 10 times, walk in the hall for 10 minute, and then return for removal of the pad. The pad was then weighed and the net weight was calculated by subtracting from the original dry weight to achieve a measure of the total urine loss during the 20 minute exercise. The pad weight was measured in grams and the accuracy of the scale was 1 gram. The positive pad weight result was defined as more than 1 gram of leakage. Each woman underwent a complete UDS before pad test, including uroflowmetry, filling (with a rate of 60mL H2O/min of 35℃ distilled water) and voiding cystometry, and stress urethral pressure profile using a two-way NO.7 French flexible Foley catheter with the SD amount in the bladder. The retest twenty-minute pad test infused with SD amount water in bladder was performed within one week after first pad test. The activities that the patients underwent were the same in test and retest 20-minute pad tests. USI was diagnosed if involuntary urine leakage was noted during filling cystometry, associated with increased intra-abdominal pressure, in the absence of a detrusor contraction. Detrusor overactivity (DO) was diagnosed if involuntary detrusor contraction occurred during filling cystometry. The exclusion criteria included no obvious USI, clinically significant urinary tract infection (UTI), and chronic pelvic inflammation. The procedures and study purpose were completely explained to the participants with fully informed consent.

A multichannel urodynamic equipment (Life-Tech, Houston, TX, USA) with computer analysis and Urovision (Urolab Janus System V, Houston, Tex) was used. All terminology conformed to the standards recommended by the ICS and Urodynamic Society. All procedures were performed by an experienced technician, and the data were interpreted by a single observer to avoid inter-observer variability.

STATA software (Version 11.0; Stata Corp, College Station, TX, USA) was used for statistical analyses. Spearman rank-correlation coefficient and intraclass correlation coefficient were tested for correlation and reliability of the test and retest results. The Wilcoxon signed rank test was tested for the difference of the test and retest. A p value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women who had fulfilled the standardization of terminology of lower urinary function from ICS were diagnosed as urodynamic stress incontinence (USI) after urodynamic study (UDS)

Exclusion Criteria:

* SUI but not USI
* Urinary tract infection
* Pelvic inflammation or malignancy
* Long term urinary catheterization

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
20-minute pad test | One week
  The pad weight or 20-minute pad test

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sutherst J, Brown M, Shawer M. Assessing the severity of urinary incontinence in women by weighing perineal pads. Lancet. 1981 May 23;1(8230):1128-30. doi: 10.1016/s0140-6736(81)92299-6. PMID 6112488
- [Background] Abrams P, Blaivas JG, Stanton SL, Andersen JT. The standardisation of terminology of lower urinary tract function. The International Continence Society Committee on Standardisation of Terminology. Scand J Urol Nephrol Suppl. 1988;114:5-19. No abstract available. PMID 3201169
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Ferreira CH, Bo K. The Pad Test for urinary incontinence in women. J Physiother. 2015 Apr;61(2):98. doi: 10.1016/j.jphys.2014.12.001. Epub 2015 Mar 3. No abstract available. PMID 25744851
- [Background] Wu WY, Sheu BC, Lin HH. Comparison of 20-minute pad test versus 1-hour pad test in women with stress urinary incontinence. Urology. 2006 Oct;68(4):764-8. doi: 10.1016/j.urology.2006.04.018. PMID 17070349
- [Background] Krhut J, Zachoval R, Smith PP, Rosier PF, Valansky L, Martan A, Zvara P. Pad weight testing in the evaluation of urinary incontinence. Neurourol Urodyn. 2014 Jun;33(5):507-10. doi: 10.1002/nau.22436. Epub 2013 Jun 24. PMID 23797972
- [Background] Lose G, Rosenkilde P, Gammelgaard J, Schroeder T. Pad-weighing test performed with standardized bladder volume. Urology. 1988 Jul;32(1):78-80. doi: 10.1016/0090-4295(88)90462-1. PMID 3388665
- [Background] Wu WY, Sheu BC, Lin HH. Twenty-minute pad test: comparison of infusion of 250 ml of water with strong-desire amount in the bladder in women with stress urinary incontinence. Eur J Obstet Gynecol Reprod Biol. 2008 Jan;136(1):121-5. doi: 10.1016/j.ejogrb.2007.02.030. Epub 2007 May 30. PMID 17540494
- [Background] Simons AM, Yoong WC, Buckland S, Moore KH. Inadequate repeatability of the one-hour pad test: the need for a new incontinence outcome measure. BJOG. 2001 Mar;108(3):315-9. doi: 10.1111/j.1471-0528.2001.00069.x. PMID 11281474